Official Title of the study: Utilizing Digital Health Approaches to Promote Early Childhood

Healthy Eating and Activity Behaviors

**NCT number** (if available): Pending **Date of the document:** January 6, 2025

#### eHEROs (Know How) Pilot Study Overview



The overall aim of the <u>e</u>lectronic <u>HE</u>althy Envi<u>RO</u>nment<u>s</u> study (eHEROs) is to transform a tested, traditional, in-person parent intervention for families of young children to a digital platform promoting healthy eating and activity behaviors and environments, and ultimately healthy growth. The intervention program is called Know-How: Building Healthy Eaters and Movers (Know-How). The intervention will be 10 weeks. Week 0 will be an introduction to the overall study followed by 9 weeks of Know How programming. *Please note that the formal name of the study is e-HEROs, but participants will only see the term Know How program/study use.* 

### **Intervention Design**

The Know-How program provides parent education on the topics of mindful parenting, healthy eating, and physical literacy and will consist of 3 components: 1) a custom mobile application (app); 2) virtual group discussions and 3) child-centered support materials mailed to participating families.

### 1. Know-How app

The Know-How app will provide parent education using a variety of modalities The 'know' will provide parents with the core information on mindful parenting, healthy eating, physical literacy and the 'how' will give strategies to incorporate the information into daily routines and activities. To facilitate the transition from the 'know' to 'how', the app with have a 'Kid Zone' will content to engage in activities with the preschooler. Content will be based on the theoretical constructs of the Adult Learning Theory and Social Cognitive Theory. Content will be divided into five modules that include A) lessons (text, audio, video), B) activities, and C) assessments.

## A. Lessons

| A. Lessons | |
|---|---|
| Table 1. Know-How Topics by Content Area | |
| Content Area | Topics |
| Mindful Parenting | Parenting Mindfully |
| | Non-Judgmental Acceptance |
| | Listening Mindfully |
| | Emotionally Mindful |
| | Parenting Compassionately |
| | Self-Regulation |
| Healthy Eating | Offering New Foods |
| | Mealtime Conversations |
| | Home Food Environment |
| Physical Literacy | Movement Skills |
| | Active Play |
| | Activity Opportunities |
| Kid Zone | Intro to the Sporks Family |
| | • Let's Eat |
| | • Let's Move |
| | • Let's Go |

#### B. Activities

To engage participants with the lesson content, activities will be interspersed within the lessons. Activities will include quizzes, goal setting and monitoring, and behavioral activities.

- Quizzes will inquire about participants:
  - Confidence in offering healthy foods, providing PA opportunities to child, engaging in positive interactions with child related to healthy eating, PA and modifying the home environment.
  - Knowledge on feeding and practices and misconceptions; physical literacy; and other core content.
- Goal Setting and monitoring activities will embed mindful parenting strategies to enactment of the 3 healthy eating topics and 3 physical literacy topics. Participants will choose at least 2 of the mindfulness prompts (watch, listen, talk, try) and plan how to practice a new behavior, record if they accomplished the plan, and reflect on the experience.
- Behavioral activities and reflections will provide participants with experiences to move from the 'know' to the 'how'. They will be asked to choose a new food to offering their child and reflect on how it went (child's sensory behaviors, liking, their experience and observations). Secondly, they will be asked to upload photos of meals and snack offerings to reflect on meal composition (which food groups were provided, portion sizes), environmental factors (who did the child eat with, mealtime environment/distractions) and timing and frequency of snacks. Related to physical activity, participants will upload short videos (15-30 seconds) of their child participating in a Kid Zone activity or practicing a movement skill. Parents will reflect on their interactions with the child (e.g., modeling, verbal encouragement, instruction, etc.).

#### C. Assessments

Two assessments will be built into the app (to complement survey distributed via REDCap) and administered at baseline and post-intervention. These assessments – Food Photography and Child Movement Skills – will require photo and video upload. To reduce participant burden of learning a new system, we have built these 2 assessments into the app.

- Food Photography: To assess mealtime food quality and intake, parents will be asked to take 2 photos of their child's meal (before the child eats (pre-meal) and post-meal) on 3 days (2 weekday and 1 weekend day) over a 7-10, day period. Along with pre-meal photo, participants will be asked to provide a text description of the meal components/ingredients. Parents will have the opportunity to provide any optional text about the meal with the post-meal photo (e.g., second servings, spilled items, an additional food item added mid meal). Photos will be downloaded and stored on
- *Child Movement Skills:* To assess movement skills, parents will be asked to record their child attempting 11 movement skills in 4 groups:
  - Locomotor 1 run, gallop slide
  - o Ball skills 1 overhand throw, underhand roll, catch
  - Locomotor 2 hop, leap, horizontal jump
  - o Ball skills 2 dribbling and kick

### 2. Group Discussions

During the 9-week intervention, participants will meet via Zoom for 6, 45-60 minute sessions to connect with a trained group facilitator (member of the research team) and a group of peers (6-8)

from their cohort. The discussions will consist of 2-3 topics (e.g., picky eating, motor development) that complement the materials from the app and allow participants to discuss their experiences, successes or challenges with the material or activities. The purpose is to build community and provide social support to the participants. Embedded within the discussions will be questions about quality of conversation (Discussions 2 & 4), acceptability of program (Discussion 3) and community belongingness (Discussion 5).

## 3. Support materials

Materials to support both assessment (e.g., balls) and programming (e.g., chef's hat and apron, activity dots, scarves, etc.) will be mailed to participants. We anticipate ~3 mailings spread out over the program. Materials are intended to support behavioral activities and to provide incentive to engage with the children's activities (KidZone) and to continue with/complete the Know How program.

| Activity | Week | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 |
| Know | Study | Introduction | | Know Your | | Know Your | | Know Your | | Summary |
| How App | Overview | | | Child | | Self | | Home | | |
| Modules | | | | | | | | | | |
| Group | 1 | | 2 | | 3 | | 4 | | 5 | 6 |
| Discussion | | | | | | | | | | |
| Support | X | | | X | | | | X | | |
| Materials | | | | | | | | | | |

**Table 2: Know How Intervention Design** 

## **Study Design**

This study is a feasibility study that will include 2 cohorts with a delayed control group (Figure 2). Study assessments will be collected at Baseline (Time 1), pre-intervention and at Post-Test (Time 2), post-intervention at the same time for both groups. No additional assessments will be collected for the delayed control group at the conclusion of implementation.



Figure 1: Study Timeline by Cohort and Intervention Group

# Measures

Table 2 outlines the measures that will be collected at either Baseline (Time 1) or Post-Intervention (Time 2). Measures will be either included in the mobile app or provided to participants via REDCap.

| <b>Activity/Testing</b> | Measures | Variables | Data Source | Time 1 2 Prior to enrollment | | IRB<br>Submission |
|---|---|---|---|---|---|---|
| Screener | Eligibility<br>Criteria | Inclusion: Participants must have a preschool-aged child (3-5 years) with no disabilities or conditions that impact typical eating and activity behaviors. Adult participants must have access to a smartphone, reliable internet at home, and can make video calls. | 0. Screener | | | |
| | | Exclusion: Adults who do not have a child aged 3-5 or child has a disability/condition. Technology access is limited. Adults who read, write or speak a language other than English. | | | | V |
| Participant<br>Information | Demographics<br>& Participant<br>Characteristics | Demographics: Age, Gender, Race, Ethnicity, Education, Income Participant Characteristics: Digital literacy, child food fussiness, physical activity ability | 1.Information Sheet | X | | <b>V</b> |
| Feasibility Primary Outcome | Recruitment | Completed interest form, eligibility status, and enrollment | Study records | X | | |
| | Retention | Proportion of intervention and app modules completers | Study records and App backend data | | X | |
| | Usability | Ease of use, complexity, confidence in using, likelihood of use | 2. Experience with Know How Program | | X | V |
| | Acceptability | Ratings of information helpfulness, goal setting, liking, willingness to recommend, desire for additional information | 2. Experience with<br>Know How Program | | X | V |
| Implementation Outcomes Primary Outcomes | Digital<br>Engagement | Delivery, receipt, and dosage - amount of time engaged by topic, features, and temporal patterns; completion rates of modules and within-app activities. | App backend data | | X | |
| | Enactment | Participation in target behaviors | Data from behavioral outcomes (below); A.Focus groups and | | X | V |

| | | | B.Interviews | | | |
|---|---|---|---|---|---|---|
| | Intention to<br>Sustain | Identify intervention strategies relating to target behaviors which were implemented or adopted | A.Focus groups and<br>B.Interviews | | X | V |
| | Peer Support | Gauge quality of conversations, sense of community as well as acceptability of programming. | 3. Group<br>Discussions | During<br>Intervention | | V |
| Behavioral Outcomes Secondary Outcomes | Mindful<br>Parenting | Listening with full attention, emotional awareness of self<br>and child, self-regulation, compassion of self and child,<br>non-judgmental acceptance of self and child | 4. Parenting | X | X | V |
| | Parenting<br>Practices | Parent-Child Feeding Practices: Autonomy (encourages exploration of new foods, offers new foods, repeatedly presents new foods) and Structure (mealtime) Physical Activity Parenting Practices: Structure (nondirective support, supportive expectation, restriction of PA inside), Autonomy (support, guided choice) Snacking Parenting Practices: Snacks to manage behavior, snack planning, monitoring, and limit setting. | 5. Child Feeding 6. Physical Activity and 7. Snacking | X | X | V |
| Outcomes Exploratory Outcomes Foo Pho Chi Mo Ski Chi Inta | Home<br>Environment | Availability of Fruit, Convenience Foods, Beverages and Whole Grains; Physical activity equipment | 8. Home Health<br>Environment | X | X | V |
| | Mealtime<br>Food<br>Photography | Mealtime food quality & intake | 9. Mealtime photos (downloaded from app) | X | X | V |
| | Child<br>Movement<br>Skills | Locomotor skills: run, gallop, hop, leap, horizontal jump, slide Ball skills: dribbling, catch, kick, overhand throw, underhand roll | 10. Movement videos (downloaded from app) | X | X | V |
| | Child Dietary<br>Intake | Frequency of child's consumption of a subset of foods – fruits, vegetables, protein, grains, beverages, dairy. | 11. Child's Diet | X | X | V |
| | Child Physical<br>Activity | Opportunities for structured and unstructured PA | 12. Physical Activity<br>Opportunities | X | X | V |

Time 1= Baseline, Time 2= Post-Intervention